CLINICAL TRIAL: NCT06291246
Title: Expediting Enrollment Into Autism-specific Intervention for Black Toddlers: A Telehealth-based Family Navigation Approach
Brief Title: Expediting Access to Services for Equity
Acronym: EASE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was prematurely terminated by funder.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-1823; K12TR004416-01 (NIH)
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Navigation (Experimental): Participants randomized to the Family Navigation condition will receive up to 4 research-based individual sessions with a trained navigator to support them in identifying and enrolling in recommended autism early intervention services. All navigation sessions will be delivered virtually via phone/Zoom.
  Interventions: Behavioral: Virtual Family Navigation
- Educational Materials (Active Comparator): The comparison condition ("Educational Materials") consists of providing the participant's caregivers information about early intervention and community-based supports (i.e., infant-toddler programs, transition to school-based supports, family support groups, local organizations. Families in this condition will receive this information throughout 4 timepoints in the first 3 months after enrolling.
  Interventions: Behavioral: Educational Materials

INTERVENTIONS:
Behavioral: Virtual Family Navigation — Participants randomized to the Family Navigation condition will receive up to 4 research-based individual sessions with a trained navigator to support them in identifying and enrolling in recommended autism early intervention services. All navigation sessions will be delivered virtually via phone/Zoom.
  Arms: Family Navigation
Behavioral: Educational Materials — The comparison condition ("Educational Materials") consists of providing the participant's caregivers information about early intervention and community-based supports (i.e., infant-toddler programs, transition to school-based supports, family support groups, local organizations. Families in this condition will receive this information throughout 4 timepoints in the first 3 months after enrolling.
  Arms: Educational Materials

SUMMARY:
The goal of this clinical trial is to assess whether telehealth-based Family Navigation (FN) expedites enrollment (e.g., reduces time in days) in community-based autism intervention for Black toddlers under the age of 4 after their initial diagnosis of autism.

The main questions it aims to answer are:

Does Family Navigation decrease the time to initiation of intervention for Black toddlers with autism?

Does Family Navigation improve developmental outcomes at 18 months post-diagnosis of autism?

Does Family Navigation improve caregiver well-being?

Caregivers in the Family Navigation condition will receive 4 research-based individual sessions with a trained navigator to support them in identifying and enrolling in recommended autism early intervention services. All navigation sessions will be delivered virtually via phone/Zoom.

Researchers will compare participants who receive family navigation to participants who receive the standard of care (educational materials) to see if family navigation outperforms the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Children up to 48 months who have a new diagnosis of autism, or who are waiting for a diagnosis of autism AND their caregiver.
* Live in Georgia or North Carolina
* Caregiver must be over the age of 18
* Their child with autism must identify as Black/African-American
* Speak conversationally fluent English.

Exclusion Criteria:

* No access to a telephone or internet connection for phone calls or video conferencing.
* Diagnosis of autism spectrum disorder is ruled out in the child.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Time to initiation of autism specific intervention | From enrollment to 6 months post.
  The date of initiation (date 1) of autism-specific intervention will be the date that families report the first session with a therapist following the diagnosis (date 2). Time will be calculated as the number of days elapsed between these two dates (date 2 - date 1).

SECONDARY OUTCOMES:
Caregiver Well-Being Score | 6 months post enrollment
  Scores on the General Well-Being Schedule will be used to measure caregiver well-being. Total scores range from 0-110. Higher scores are indicative of more positive well-being. There are 3 proposed scoring cut-points: 0-60 reflects "severe distress", 61-72 reflects "moderate distress", and 73-110 reflects "positive well-being).
Child's Developmental Functioning Score | 18 months post enrollment
  The Early Learning Composite from the Mullen Scales of Early Learning (MSEL) will be used to measure developmental functioning. The Early Learning Composite (ELC) is a standardized composite score derived from the 5 subtests measured on the MSEL. It has a mean of 100 and a standard deviation of 15. Higher scores indicate stronger performance.
Child's Adaptive Functioning Score | 18 months post enrollment
  The Adaptive Behavior Assessment Scale, Third Edition (ABAS-3) will be used to measure adaptive functioning. The ABAS-3 assesses 3 domains of adaptive behavior, including Conceptual, Social, and Practical. The General Adaptive Composite (GAC) is a composite score derived from the 4 domains. It has a mean of 100 and a standard deviation of 15. Higher scores indicate stronger adaptive behavior skills.
Appropriateness of Intervention Score | 6 months after enrollment
  The Intervention Appropriateness Measure (IAM) is a 4 question survey that assesses a participant's experience with or thoughts about the intervention's appropriateness. A scaled score can be created by averaging the item-level responses. Scaled score values range from 1 to 5. Cut-off scores or norms for interpretation are not yet available; however, higher scores indicate greater appropriateness.
Feasibility of Intervention Score | 6 months after enrollment
  The Feasibility of Intervention Measure (FIM) is a 4 question survey that assesses a participant's experience with or thoughts about the intervention's feasibility. A scaled score can be created by averaging the item-level responses. Scaled score values range from 1 to 5. Cut-off scores or norms for interpretation are not yet available; however, higher scores indicate greater appropriateness.
Acceptability of Intervention Score | 6 months after enrollment
  The Acceptability of Intervention Measure (AIM) is a 4 question survey that assesses a participant's experience with or thoughts about the intervention's acceptability. A scaled score can be created by averaging the item-level responses. Scaled score values range from 1 to 5. Cut-off scores or norms for interpretation are not yet available; however, higher scores indicate greater appropriateness.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Caravella, PhD, Principal Investigator — UNC
Locations (1):
- Carolina Institute for Developmental Disabilities, Carrboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 9 to 36 months following publication.
Access Criteria: Investigator must have approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

DOCUMENTS (1):
  • Informed Consent Form (2025-02-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT06291246/ICF_000.pdf